CLINICAL TRIAL: NCT05508308
Title: Automated Oxygen Control for Preterm Infants On Continuous Positive Airway Pressure (CPAP): Phase 1/2 Trial In Southwest Nigeria
Brief Title: Automated Versus Manual Control Of Oxygen For Preterm Infants On Continuous Positive Airway Pressure In Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: University of Tasmania (Other); University College Hospital, Ibadan (Other); Sacred Heart Hospital Lantoro (Unknown); University of Ibadan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HREC84704
Record Dates: First submitted 2022-08-12; First posted 2022-08-19 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Neonatal Respiratory Distress Related Conditions; Neonatal Respiratory Failure; Prematurity; Oxygen Toxicity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Preterm infants on bCPAP are managed with each mode of oxygen control for 24 hours, prior to crossing over to the other mode of control. Change over simply involves flicking the computer switch from manual to automated control (or vice versa) and it is enacted immediately. It does not require any adjustment or interruption of the CPAP and it does not involve additional action from clinical staff. While the fraction of inspired oxygen (FiO2) adjustments have their effect relatively rapidly, we will apply a 1 h washout period (dropping this data from analysis) to avoid contamination between arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual oxygen control (Active Comparator): Oxygen therapy delivered with bCPAP as per standard practice, except for the addition of continuous pulse oximetry. Nursing staff will make manual adjustments to Fraction of Inspired Oxygen (FiO2) provided to infants on bCPAP. Oxygen saturations (SpO2) will be monitored by continuous pulse oximetry, and nurses asked to target the range of SpO2 91-95%. Pulse oximeter alarms will be set to alert nurses to periods of hypoxaemia (SpO2<88%) and hyperoxaemia (SpO2>96%).
  Interventions: Other: Manual oxygen control
- OxyMate Automated Oxygen Control (Experimental): Automated control of oxygen therapy partnered with bCPAP delivered as per standard practice. The automated oxygen control set-up (OxyMate) will consist of: continuous pulse oximetry input, a computer algorithm (VDL1.1) that calculates changes to delivered FiO2 based on the input SpO2, and a mechanism to automatically effect changes to delivered FiO2. The system will target an SpO2 of 93% (mid-point of the target range). There will be several embedded safety mechanisms, including the ability to manually over-ride OxyMate at any stage. Pulse oximeter alarms will be as for the manual control arm, with additional automated system alarms in place.
  Interventions: Device: OxyMate

INTERVENTIONS:
Device: OxyMate — Automated Oxygen Control algorithm (VDL 1.1) coupled with Diamedica Baby CPAP device
  Arms: OxyMate Automated Oxygen Control
Other: Manual oxygen control — Guidelines and training in FiO2 titration to achieve a target range of SpO2. Health workers instructed in responding to continuous pulse oximetry readings and alarms
  Arms: Manual oxygen control

SUMMARY:
One in ten babies are born preterm (<37 weeks gestation) globally. Complications of prematurity are the leading cause of death in children under 5 years, with the highest mortality rate in Sub-Saharan Africa (SSA). Low flow oxygen, and respiratory support - where an oxygen/air mixture is delivered under pressure - are life saving therapies for these babies. Bubble Continuous Positive Airway Pressure (bCPAP) is the mainstay of neonatal respiratory support in SSA.

Oxygen in excess can damage the immature eyes (Retinopathy of Prematurity [ROP]) and lungs (Chronic Lung Disease) of preterm babies. Historically, in well-resourced settings, excessive oxygen administration to newborns has been associated with 'epidemics' of ROP associated blindness. Today, with increasing survival of preterm babies in SSA, and increasing access to oxygen and bCPAP, there are concerns about an emerging epidemic of ROP. Manually adjusting the amount of oxygen provided to an infant on bCPAP is difficult, and fearing the risks of hypoxaemia (low oxygen levels) busy health workers often accept hyperoxaemia (excessive oxygen levels). Some well resourced neonatal intensive care units globally have adopted Automated Oxygen Control (AOC), where a computer uses a baby's oxygen saturation by pulse oximetry (SpO2) to frequently adjust how much oxygen is provided, targetting a safe SpO2 range. This technology has never been tested in SSA, or partnered with bCPAP devices that would be more appropriate for SSA.

This study aims to compare AOC coupled with a low cost and robust bCPAP device (Diamedica Baby CPAP) - OxyMate - with manual control of oxygen for preterm babies on bCPAP in two hospitals in south west Nigeria. The hypothesis is that OxyMate can significantly and safely increase the proportion of time preterm infants on bCPAP spend in safe oxygen saturation levels.

DETAILED DESCRIPTION:
Trial description: A randomised cross-over trial of manual versus automated control of oxygen (OxyMate) for preterm infants on bCPAP. This trial will use an established technology (automated oxygen titration algorithm, VDL1.1) partnered with a low-cost bCPAP device in a low-resource setting. It will involve preterm infants requiring bCPAP respiratory support with allocation to OxyMate or manual oxygen control for consecutive 24 h periods in random sequence.

Objectives: This trial seeks to examine safety and potential efficacy of our automated oxygen configuration (OxyMate) in preterm infants in a setting characterised by financial constraints, workforce limitations, and underdeveloped infrastructure, and assess contextual feasibility and appropriateness to inform future definitive clinical trials and product development.

ELIGIBILITY:
Inclusion Criteria:

* <34 weeks gestation (or birth weight < 2kg if gestation not known)
* ≥12 hours old
* Receiving CPAP support and supplemental oxygen (FiO2 >0.21) for respiratory insufficiency
* Projected requirement for CPAP and oxygen therapy for > 48 hours

Exclusion Criteria:

* Deemed likely to fail CPAP in the next 48 hours
* Deemed clinically unstable or recommended for palliation by treating team
* Cause of hypoxaemia likely to be non-respiratory - e.g. cyanotic heart disease
* Informed consent from parent/guardians not obtained

Ages: 12 Hours to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Proportion of time in target SpO2 range | Measured for each 24 hour study epoch
  Proportion of time (over total recorded time) in the target SpO2 range (91-95%, or 91-100% when in room air). Measured as %time

SECONDARY OUTCOMES:
Proportion of time in target SpO2 range when receiving supplemental oxygen | Measured for each 24 hour study epoch
  Proportion of time (over total recorded time) in SpO2 target range (91-95%) when receiving supplemental oxygen. Measured as %time when receiving oxygen
Proportion of time in hypoxaemia | Measured for each 24 hour study epoch
  Proportion of time (over total recorded time) with SpO2<90% (hypoxaemia). Measured as %time
Proportion of time in severe hypoxaemia | Measured for each 24 hour study epoch
  Proportion of time (over total recorded time) with SpO2 <80% (severe hypoxaemia). Measured as %time
Frequency of prolonged hypoxaemia episodes | Measured for each 24 hour study epoch
  Frequency of 30 seconds episodes with SpO2 continuously <80% (severe hypoxaemic episodes). Measured as episodes per hour
Proportion of time in hyperoxaemia | Measured for each 24 hour study epoch
  Proportion of time (over total recorded time) with SpO2 >96% when receiving supplemental oxygen (hyperoxaemia). Measured as %time when receiving oxygen
Proportion of time in severe hyperoxaemia | Measured for each 24 hour study epoch
  Proportion of time (over total recorded time) with SpO2 >98% when receiving supplemental oxygen (severe hyperoxaemia). Measured as %time when receiving oxygen
Frequency of prolonged hyperoxaemia episodes | Measured for each 24 hour study epoch
  Frequency of 30 seconds episodes with SpO2 continuously >96% (hyperoxaemic episodes). Measured as episodes per hour
Manual FiO2 adjustments | Measured for each 24 hour study epoch
  Frequency of manual FiO2 adjustments. Measured as FiO2 adjustments/hour
No response to prolonged severe hypoxaemia (frequency) | Measured for each 24 hour study epoch
  Number of periods of no FiO2 increment for ≥30 seconds with SpO2 <80% (i.e. failure to respond to severe hypoxaemia). Measured as episodes per hour
No response to prolonged severe hypoxaemia (duration) | Measured for each 24 hour study epoch
  Duration of periods of no FiO2 increment for ≥30 seconds with SpO2 <80% (i.e. failure to respond to severe hypoxaemia). Measured as mean duration per episode
Severe hypoxaemia with bradycardia (frequency) | Measured for each 24 hour study epoch
  Number of periods with SpO2 <80% for ≥30 seconds with any bradycardia (heart rate <100 bpm). Measured as episodes per hour
Severe hypoxaemia with bradycardia (duration) | Measured for each 24 hour study epoch
  Duration of periods with SpO2 <80% for ≥30 seconds with any bradycardia (heart rate <100 bpm). Measured as mean duration per episode
Device malfunction | Measured through to OxyMate study completion: estimated 20 weeks
  Number of OxyMate malfunction events
Acceptability and usability | Completed for each participant (health workers) at end of an infant's study period (49 hours). Results recorded for unique health workers through to OxyMate study completion: estimated 20 weeks
  Mean/median user acceptability score (total and per question) on Likert scale from structured questionnaire. Scores range from 1 (strongly disagree) to 5 (strongly agree) with posed statement or question
Costs | Measured at completion of OxyMate study: an estimated 20 weeks
  Total costs of prototype system (Diamedica +/- Automated Oxygen control - OxyMate)
Duration of CPAP and oxygen therapy | Completed for each participant at end of their study period: 49 hours from study commencement
  Duration of time on CPAP with supplemental oxygen. Measured in hours
CPAP in room air | Completed for each participant at end of their study period: 49 hours from study commencement
  Duration of time on CPAP in room air. Measured in hours
Time on low flow oxygen | Completed for each participant at end of their study period: 49 hours from study commencement
  Duration of time on low-flow oxygen therapy. Measured in hours
Final discharge outcome | Up to 4 weeks post enrollment
  Measured as categorical outcome (died in hospital, discharged well, discharged against medical advice, other)
Length of stay | Up to 4 weeks post enrollment
  Measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Hamish R Graham, PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (2):
- Nigeria (2):
  - Sacred Heart Hospital, Lantoro, Abeokuta
  - University College Hospital, Agodi, Ibadan

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for the final analysis of the OxyMate trial will be available two months after publication of the primary outcome.
  Documents that will be made available are Study Protocol and Informed Consent Form. Data may be obtained from the Murdoch Children's Research Institute (MCRI) by emailing hamish.graham@mcri.edu.au and mctc@mcri.edu.au
Supporting Information: Study Protocol, ICF
Time Frame: 2 months after publication of the primary outcome.
Access Criteria: Prior to releasing any data the following are required:
  1. A Data Transfer Agreement must be signed between relevant parties.
  2. The MCRI Sponsorship Committee must review and approve your protocol and statistical analysis plan which must include and describe how the data will be used and analysed.
  3. An Authorship Agreement must be agreed to and signed between relevant parties. The Agreement must include details regarding appropriate recognition. Authorship may not be justifiable but some form of acknowledgment is requested.
  4. Agreement to cover any additional costs relating to the provision of the data.
  5. Evidence of ethics approval or waiver of approval, to be compliant with the data transfer agreement and ethics requirement at MCRI.
  Data will only be shared with a recognised research institution where the MCRI Sponsorship Committee has approved the proposed analysis plan.

REFERENCES:
- [Result] Chawanpaiboon S, Vogel JP, Moller AB, Lumbiganon P, Petzold M, Hogan D, Landoulsi S, Jampathong N, Kongwattanakul K, Laopaiboon M, Lewis C, Rattanakanokchai S, Teng DN, Thinkhamrop J, Watananirun K, Zhang J, Zhou W, Gulmezoglu AM. Global, regional, and national estimates of levels of preterm birth in 2014: a systematic review and modelling analysis. Lancet Glob Health. 2019 Jan;7(1):e37-e46. doi: 10.1016/S2214-109X(18)30451-0. Epub 2018 Oct 30. PMID 30389451
- [Result] WHO Recommendations on Interventions to Improve Preterm Birth Outcomes. Geneva: World Health Organization; 2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK321160/ PMID 26447264
- [Result] Gilbert C. Retinopathy of prematurity: a global perspective of the epidemics, population of babies at risk and implications for control. Early Hum Dev. 2008 Feb;84(2):77-82. doi: 10.1016/j.earlhumdev.2007.11.009. Epub 2008 Jan 29. PMID 18234457
- [Result] BOOST-II Australia and United Kingdom Collaborative Groups; Tarnow-Mordi W, Stenson B, Kirby A, Juszczak E, Donoghoe M, Deshpande S, Morley C, King A, Doyle LW, Fleck BW, Davis PG, Halliday HL, Hague W, Cairns P, Darlow BA, Fielder AR, Gebski V, Marlow N, Simmer K, Tin W, Ghadge A, Williams C, Keech A, Wardle SP, Kecskes Z, Kluckow M, Gole G, Evans N, Malcolm G, Luig M, Wright I, Stack J, Tan K, Pritchard M, Gray PH, Morris S, Headley B, Dargaville P, Simes RJ, Brocklehurst P. Outcomes of Two Trials of Oxygen-Saturation Targets in Preterm Infants. N Engl J Med. 2016 Feb 25;374(8):749-60. doi: 10.1056/NEJMoa1514212. Epub 2016 Feb 10. PMID 26863265
- [Result] Askie LM, Darlow BA, Finer N, Schmidt B, Stenson B, Tarnow-Mordi W, Davis PG, Carlo WA, Brocklehurst P, Davies LC, Das A, Rich W, Gantz MG, Roberts RS, Whyte RK, Costantini L, Poets C, Asztalos E, Battin M, Halliday HL, Marlow N, Tin W, King A, Juszczak E, Morley CJ, Doyle LW, Gebski V, Hunter KE, Simes RJ; Neonatal Oxygenation Prospective Meta-analysis (NeOProM) Collaboration. Association Between Oxygen Saturation Targeting and Death or Disability in Extremely Preterm Infants in the Neonatal Oxygenation Prospective Meta-analysis Collaboration. JAMA. 2018 Jun 5;319(21):2190-2201. doi: 10.1001/jama.2018.5725. PMID 29872859
- [Result] Sink DW, Hope SA, Hagadorn JI. Nurse:patient ratio and achievement of oxygen saturation goals in premature infants. Arch Dis Child Fetal Neonatal Ed. 2011 Mar;96(2):F93-8. doi: 10.1136/adc.2009.178616. Epub 2010 Oct 30. PMID 21037284
- [Result] Gantz MG, Carlo WA, Finer NN, Rich W, Faix RG, Yoder BA, Walsh MC, Newman NS, Laptook A, Schibler K, Das A, Higgins RD; SUPPORT Study Group of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Achieved oxygen saturations and retinopathy of prematurity in extreme preterms. Arch Dis Child Fetal Neonatal Ed. 2020 Mar;105(2):138-144. doi: 10.1136/archdischild-2018-316464. Epub 2019 Jun 22. PMID 31229956
- [Result] Hagadorn JI, Furey AM, Nghiem TH, Schmid CH, Phelps DL, Pillers DA, Cole CH; AVIOx Study Group. Achieved versus intended pulse oximeter saturation in infants born less than 28 weeks' gestation: the AVIOx study. Pediatrics. 2006 Oct;118(4):1574-82. doi: 10.1542/peds.2005-0413. PMID 17015549
- [Result] Walker PJB, Bakare AA, Ayede AI, Oluwafemi RO, Olubosede OA, Olafimihan IV, Tan K, Duke T, Falade AG, Graham H. Using intermittent pulse oximetry to guide neonatal oxygen therapy in a low-resource context. Arch Dis Child Fetal Neonatal Ed. 2020 May;105(3):316-321. doi: 10.1136/archdischild-2019-317630. Epub 2019 Aug 28. PMID 31462405
- [Result] Sturrock S, Williams E, Dassios T, Greenough A. Closed loop automated oxygen control in neonates-A review. Acta Paediatr. 2020 May;109(5):914-922. doi: 10.1111/apa.15089. Epub 2019 Nov 27. PMID 31715041
- [Result] Mitra S, Singh B, El-Naggar W, McMillan DD. Automated versus manual control of inspired oxygen to target oxygen saturation in preterm infants: a systematic review and meta-analysis. J Perinatol. 2018 Apr;38(4):351-360. doi: 10.1038/s41372-017-0037-z. Epub 2018 Jan 2. PMID 29296004
- [Result] Dargaville PA, Marshall AP, McLeod L, Salverda HH, Te Pas AB, Gale TJ. Automation of oxygen titration in preterm infants: Current evidence and future challenges. Early Hum Dev. 2021 Nov;162:105462. doi: 10.1016/j.earlhumdev.2021.105462. Epub 2021 Sep 4. PMID 34511288
- [Result] Salverda HH, Cramer SJE, Witlox RSGM, Gale TJ, Dargaville PA, Pauws SC, Te Pas AB. Comparison of two devices for automated oxygen control in preterm infants: a randomised crossover trial. Arch Dis Child Fetal Neonatal Ed. 2022 Jan;107(1):20-25. doi: 10.1136/archdischild-2020-321387. Epub 2021 Jun 10. PMID 34112721
- [Result] Plottier GK, Wheeler KI, Ali SK, Fathabadi OS, Jayakar R, Gale TJ, Dargaville PA. Clinical evaluation of a novel adaptive algorithm for automated control of oxygen therapy in preterm infants on non-invasive respiratory support. Arch Dis Child Fetal Neonatal Ed. 2017 Jan;102(1):F37-F43. doi: 10.1136/archdischild-2016-310647. Epub 2016 Aug 29. PMID 27573518
- [Result] Dargaville PA, Sadeghi Fathabadi O, Plottier GK, Lim K, Wheeler KI, Jayakar R, Gale TJ. Development and preclinical testing of an adaptive algorithm for automated control of inspired oxygen in the preterm infant. Arch Dis Child Fetal Neonatal Ed. 2017 Jan;102(1):F31-F36. doi: 10.1136/archdischild-2016-310650. Epub 2016 Sep 15. PMID 27634820
- [Result] Dargaville PA, Marshall AP, Ladlow OJ, Bannink C, Jayakar R, Eastwood-Sutherland C, Lim K, Ali SKM, Gale TJ. Automated control of oxygen titration in preterm infants on non-invasive respiratory support. Arch Dis Child Fetal Neonatal Ed. 2022 Jan;107(1):39-44. doi: 10.1136/archdischild-2020-321538. Epub 2021 May 7. PMID 33963005
- [Derived] Subhi R, McLeod L, Ayede AI, Dedeke IO, Risikat Q, Akanbi AR, Fasasi AB, Bakare AA, Adeniyi OH, Akinrinoye O, Adeigbe O, Dargaville GF, Walker P, Grobler AC, Mosebolatan O, Badurdeen S, Gale TJ, Falade AG, Dargaville PA, Graham HR. Automated oxygen control for preterm infants receiving continuous positive airway pressure in southwest Nigeria: an open-label, randomised, crossover trial. Lancet Glob Health. 2025 Feb;13(2):e246-e255. doi: 10.1016/S2214-109X(24)00458-3. PMID 39890225